CLINICAL TRIAL: NCT02462239
Title: Impact of Positron Emission Tomography (PET) Imaging in Muscle-invasive Urothelial Carcinoma of the Bladder Staging
Acronym: PET MUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Cancer Care Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2013-PETMUSE
Record Dates: First submitted 2015-05-27; First posted 2015-06-04 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Muscle-invasive Bladder Cancer
Keywords: Muscle-invasive bladder cancer; Bladder cancer; PET imaging; FDG
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole-body FDG PET-CT (Experimental): Whole-body FDG PET-CT (Experimental arm)
  Interventions: Other: Whole-body FDG PET-CT
- No PET-CT (No Intervention): No PET-CT (Control arm)

INTERVENTIONS:
Other: Whole-body FDG PET-CT
  Other Names: PET-CT imaging
  Arms: Whole-body FDG PET-CT

SUMMARY:
Bladder cancer is the fifth most common cancer in Canada and there has been relatively little progress in altering its clinical course over the last three decades. One of the major problems identified in the management of this disease, is under staging of muscle invasive disease which can lead to suboptimal treatment and outcomes. PET-CT has the potential to more accurately stage MIBC than standard CT by detecting pelvic adenopathy and/or distant sites of disease that may not be found on standard imaging. In the former situation, more aggressive therapy with extended lymph node dissection and/or neoadjuvant chemotherapy prior to cystectomy can be offered. While in the latter situation patients can be spared the morbidity of a cystectomy performed in a setting of metastatic disease. This study will address whether PET-CT adds a clinically meaningful difference in care.

DETAILED DESCRIPTION:
A multicenter randomized controlled trial will be performed. Patients usually present with symptoms (e.g., painless hematuria). The urologist will perform cystoscopy and if urothelial cancer of the bladder is suspected, the patient is taken to the operating room for an examination under anesthesia (EUA) and a TURBT. If this shows muscle invasion then conventional staging with CT chest, abdomen, and pelvis is performed. The patient who has TNM Stage T2a-T4a N0-3 M0 is eligible to be enrolled in the trial. Eligible consenting patients will be randomized 2:1 to PET-CT or none (Control). The actual treatment received by the patient will be documented. The primary outcome measure is treatment received.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with newly diagnosed muscle-invasive high grade urothelial carcinoma of the bladder (TNM stage T2a-T4a, N0-3, M0), who are eligible for either radical cystectomy or radiotherapy-based bladder conservation.
* Being considered for treatment of curative intent.

Exclusion Criteria:

* Age < 18 years.
* ECOG performance status >2.
* Predominant histology (>50% of specimen) involves non-urothelial cell carcinoma.
* Prior partial cystectomy.
* Prior pelvis surgery that obviates a completed extended lymphadenectomy (e.g., aorto-femoral/iliac bypass) or for whom the surgeon feels that their ability to perform a standard or extended pelvic node dissection would be compromised.
* Contraindications to FDG PET-CT.
* Inability to lie supine for imaging with PET-CT.
* Inadequate hepatic function:

  (i) Bilirubin >1.5 X ULN and (ii) SGOT and Alkaline phosphatase >3 X ULN
* History of another invasive malignancy within the previous 5 years with the exception of non-melanoma skin cancer.
* Known pregnancy or lactating female.
* Inability to complete the study or required follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Treatment received | 5 years
  For patients with planned cystectomy, treatment received includes: avoidance of planned cystectomy and node dissection, an extended (vs standard) node dissection (or standard dissection when extended is the surgeon's usual practice), use of neoadjuvant chemotherapy (vs no neoadjuvant chemotherapy). For patients with planned bladder conservation, treatment received includes: avoidance of bladder and nodal radiation (vs bladder only or no radiation) and use of neoadjuvant chemotherapy (or not).

SECONDARY OUTCOMES:
Disease-free survival | 5 years
  Disease-free survival defined as objectively defined (RECIST criteria, version 1.1.) local or distant recurrence or death.
Overall survival | 5 years
  Overall survival defined by all-cause mortality.
Quality of life analysis | 5 years
  Overall QOL assessed using the EORTC QLQ-C30 version 3.
Health economic analysis | 5 years
  Health economic analysis assessed using EQ-5D health utility questionnaire and total healthcare costs.

OTHER OUTCOMES:
Change in planned management | 5 years
  Assess change in planned management with actual treatment delivered in both pre-operative PET-CT versus no PET-CT (control) patients.
Clinical and pathology response to chemotherapy using interim response of FDG PET-CT after 2 cycles of chemotherapy | 5 years
  Explore if interim response on FDG PET-CT after 2 cycles of chemotherapy is associated with clinical and pathology response to chemotherapy and if early interim metabolic response correlates with other outcome measures including DFS and OS.

CONTACTS AND LOCATIONS:
Overall Officials: Srikala Sridhar, MD, Principal Investigator — Princess Margaret Hospital, Canada; Nicholas Power, MD, Principal Investigator — LHSC-Victoria Hospital; Som Mukherjee, MD, Principal Investigator — Juravinski Cancer Centre; Ur Metser, MD, Principal Investigator — Princess Margaret Hospital, Canada; Mark Levine, MD, Study Director — Ontario Clinical Oncology Group (OCOG)
Locations (6):
- Canada (6):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No